CLINICAL TRIAL: NCT01519362
Title: A Woman Suffered From Leukocytopenia and Widespread Migration After Polyacrylamide Hydrogel (PAAG) Injection in Epicranial Aponeurosis
Status: Completed | Type: Observational
Sponsor: Duo Zhang (Other)
Responsible Party: Sponsor-Investigator, Duo Zhang, professor, The First Hospital of Jilin University
Organization: The First Hospital of Jilin University (Other)
Other Study IDs: zhangduo
Record Dates: First submitted 2012-01-24; First posted 2012-01-26 (Estimated); Last update posted 2012-01-26 (Estimated); Status verified 2012-01

CONDITIONS: Complication
Keywords: Polyacrylamide hydrogel; leukocytopenia; migration; complication; epicranial aponeurosis; PAAG injection
MeSH Terms: conditions — Leukopenia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Polyacrylamide hydrogel (PAAG) has been used as an injectable filler for soft tissue augmentation in different parts of the body , such as face, breast , or even penis for more than a decade . However, there are never reports about the application of a large amount of PAAG in epicranial aponeurosis to change the contour of the upper cranium accompanied with leukocytopenia. This fancy application turned out to be a disaster for the women who suffered from leukocytopenia , widespread migration of PAAG, recurrent swelling of the affected tissues and temporal pain changing with the temperature and the facial expression .

ELIGIBILITY:
Inclusion Criteria:

* PAAG injected into bilateral temporal epicranial aponeurosis

Exclusion Criteria:

* PAAG injected into other parts of the body

Ages: 50 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: A 50-year-old lady had PAAG injected into her bilateral temporal epicranial aponeurosis for augmentation
Sampling Method: Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2011-10